CLINICAL TRIAL: NCT03071939
Title: Pilot Study of a New Insight Assessment Tool
Brief Title: Cognate Patient Care Insight Scale
Acronym: EIPSP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the investigator left our institution
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-A01716-45
Record Dates: First submitted 2017-02-28; First posted 2017-03-07 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: One arm in this study comprising 119 patients and one of their relatives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with schizophrenia and their designated relatives (Other): Evaluation of the patient's insight (an inclusion phase, followed by two evaluation phases on D0 and D7) by the patient, his / her close and two caregivers (inter-judicial fidelity)
  Interventions: Other: Assessment of the insight of schizophrenic patients by themselves, their relatives and caregivers

INTERVENTIONS:
Other: Assessment of the insight of schizophrenic patients by themselves, their relatives and caregivers — This study will evaluate the insight of the patient, something carried out in common practice within the Eastern Pole (CH Le Vinatier). This assessment will take place in the specific services where patients are cared for. It will make it possible to evaluate insight more closely by comparing the opinions of the three actors. There is no risk in this study.
  The study will be carried out over 2 years with a recruitment of 119 patients responding to the diagnosis of schizophrenia, taken care of within the Eastern Pole (Intra and Extrahospital services).

SUMMARY:
Schizophrenia is a disease of young adults that affects 1% of the general population. According to numerous studies, it has been estimated that between 50% and 80% of patients with schizophrenia do not consider to have a mental disorder and are therefore not aware of their disorders. A poor degree of insight is associated with poor compliance, a higher number of re-hospitalizations, altered social and relational functioning, and a higher number of suicides and violent behaviors. This is why insight, which is an essential dimension of psychopathology, must be evaluated, as it depends to a large extent on the therapeutic alliance, adherence to treatment, likelihood of relapse and prognosis.

DETAILED DESCRIPTION:
Evaluation (test, re-test) This new tool for assessing insight will allow for a discrepancy in assessment and a more refined assessment with a view to developing specific care for the patient and / or the relative with regard to the three dimensions Evaluated: disease, treatment and functional implications

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* Age from 18 to 50 years old
* Stabilized clinical condition (without therapeutic modification during the month prior to inclusion)
* French language read, spoken and understood (patient and family member)
* Having given his consent
* Agreement of the guardian for persons under guardianship
* Consent of the relative

Exclusion Criteria:

* Refusal of patient or legal guardian
* Refusal of the loved one
* Patient and / or neurological disorder of neurological origin of vascular, infectious or neurodegenerative origin

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-02 (Estimated); Primary Completion 2020-01-02 (Estimated); Study Completion 2020-04-02 (Estimated)

PRIMARY OUTCOMES:
Concurrent validity of the hetero-evaluation scale by studying its correlation with the results obtained, for the same persons, on the SUMD scale (Scale to Assess Unawareness of Mental Disorder) | two years
  Correlation higher than 0.40 in the Bravais-Pearson test between the caregiver's hetero-evaluation scale and the Scale to Assess Understanding of Mental Disorder (SUMD)

SECONDARY OUTCOMES:
Correlation greater than 0.40 to inter-judge fidelity to Cohen's Kappa test | two years
  Inter-judicial fidelity will be measured with Cohen's Kappa test, which is a coefficient to measure the agreement between two qualitative variables with the same modalities. Conventionally, it is used to measure the degree of concordance between the stages Awarded by two judges. It can also be applied to measure an intra-observer agreement.
  The closer the ratio is to 1, the closer the gap between the observed chord proportion and the theoretical proportion of "random" chords approaches the gap between the perfect tuning of the two observers and their random match. The coefficient is always between -1 and 1 (maximum agreement).
Cronbach's alpha coefficient with a value of 0.7 measuring internal consistency | two years
  Internal consistency will be measured with the Cronbach alpha coefficient, sometimes referred to simply as the coefficient.
  Which is a statistic used especially in psychometrics to measure the internal consistency (or reliability) of the questions asked during a test (the answers to the questions on the same subject to be correlated). Its value is between 0 and 1, being considered "acceptable" from 0.7. It therefore allows estimation of the fidelity of the score to a test.
Correlation greater than 0.40 at the Bravais-Pearson test measuring test fidelity, re-testing | two years
  This coefficient makes it possible to detect the presence or absence of a linear relationship between two continuous quantitative characters. To calculate this coefficient, one must first calculate the covariance. Covariance is the mean of the product of deviations from the mean. The linear correlation coefficient of two characters X and Y is equal to the covariance of X and Y divided by the product of the standard deviations of X and Y. It can be shown that this coefficient varies between -1 and +1

CONTACTS AND LOCATIONS:
Overall Officials: MAGES Nicolas, MDPH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No